CLINICAL TRIAL: NCT00175357
Title: North American Opiate Medication Initiative (NAOMI): Multi-Centre, Randomized Controlled Trial of Heroin-Assisted Therapy for Treatment-Refractory Injection Opiate Users
Brief Title: NAOMI: A Study to Compare Medically-prescribed Heroin With Oral Methadone in Chronic Opiate Addiction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P99-0209; 03-2316
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2014-09-29 (Estimated); Status verified 2014-09

CONDITIONS: Opiate Addiction
Keywords: Opiate addiction; medical heroin; methadoneRCT
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Methadone; Heroin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Oral methadone
  Interventions: Drug: Methadone
- 2 (Experimental): Injected diacetylmorphine
  Interventions: Drug: Diamorphine hydrochloride

INTERVENTIONS:
Drug: Methadone — The dose of the drug will be determined by a physician. The oral drug will be administered 1 dose per days, 7 days per week.
  Arms: 1
Drug: Diamorphine hydrochloride — The dose of the drug will be determined by a physician. The injected drug will be administered up to 3 doses per day, 7 days per week.
  Arms: 2

SUMMARY:
The objective of this study is to determine whether the closely supervised provision of injectable, pharmaceutical-grade heroin (in combination with oral methadone) is more effective than methadone therapy alone in recruiting, retaining, and benefiting long-term heroin users who have not been helped by current standard treatment options.

DETAILED DESCRIPTION:
This is a two-centre (Vancouver, Montreal) RCT involving a total of 235 volunteers. Eligible participants will be randomized to injectable heroin combined with oral methadone as desired (45%) versus oral methadone alone (45%). A subset of 10% will be randomized to injectable hydromorphone (Dilaudid™). Hydromorphone and heroin will be given in a double-blind fashion; the purpose is to permit validation of reported illicit use of heroin through urine testing in the hydromorphone group. Research visits will be conducted quarterly and will occur independently of treatment clinic visits. Incentives will be used to maintain research follow-up whether or not the subject is retained in treatment. The analysis will be under intent-to-treat. The primary outcomes of interest are 1) recruitment and retention in the study and 2) illicit drug use and criminal behavior (as determined by the Europ-ASI) at 12 months. Secondary outcomes are measures of social function (e.g., social integration and functioning, quality of life) and cost-benefit/effectiveness of the interventions.

ELIGIBILITY:
Inclusion Criteria:

1. Opioid Dependence as confirmed by DSM-IV diagnostic criteria
2. 25 years of age or older
3. 5 years or more of opioid use
4. Regular opioid injection use in the past month and in at least 8 months in the past 12 months (self reported; regular use - defined as injecting opioids for at least 4 days or more in a week); 50% or more of the injections during the prior year must have involved heroin).
5. Minimum of one-year residence in site/city location
6. No enrollment in any other opioid substitution (e.g. methadone) program within the prior 6 months - enrollment is defined as having received at least 45 milligrams of prescribed methadone per day on any 30 consecutive days or more in the prior 6 months
7. At least two previous episodes of opiate addiction treatment (methadone maintenance, detoxification, residential care, etc) during which, on at least one occasion, the patient received at least 60 mg of methadone daily for at least 30 days in a 40 day period
8. Willingness and ability to adhere to study protocol and follow-up schedule as determined through the three-week pre-randomization period (see Section C.4)
9. Documentation of fulfillment of the above study criteria (prison records, treatment records, cohort study enrollment, urine sampling)
10. Provide written and informed consent.

Exclusion Criteria:

1. Diagnosis of severe medical or psychiatric conditions that are contra-indicated for heroin treatment
2. Pregnancy upon study entry
3. On parole or with current justice system involvement that is likely to result in an extended period of incarceration (more than 4 months) during the study period (e.g. scheduled trial for an indictable offense, jail, etc)
4. Hydromorphone is a class C teratogen and should not be given to pregnant women. All female subjects upon study entry will be urged to engage only in protected sexual intercourse and will provide consent to undergo monthly pregnancy tests during the course of the study.
5. Serum bilirubin >2.5 x normal
6. Stage II or greater hepatic encephalopathy
7. Chronic respiratory disease resulting in resting respiratory rate >20/minute
8. Bipolar Mood Disorder, Schizophrenia or other psychotic disorder with active psychotic symptoms within the past 6 months
9. Major Depression refractory to medical management or requiring electroconvulsive therapy within the past 12 months.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2005-03; Primary Completion 2007-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Recruitment and retention in the study at 12 months | 12 months
Illicit drug use and criminal behavior at 12 months. | 12 months

SECONDARY OUTCOMES:
social integration, functioning, quality of life at 12 and 24 months; and cost-effectiveness at 12 months | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Martin T Schechter, MD, PhD, Principal Investigator — University of British Columbia
Locations (2):
- Canada (2):
  - University of British Columbia Faculty of Medicine, Vancouver, British Columbia
  - University of Montreal, Montreal, Quebec

REFERENCES:
- [Derived] Oviedo-Joekes E, Marchand K, Lock K, Chettiar J, Marsh DC, Brissette S, Anis AH, Schechter MT. A chance to stop and breathe: participants' experiences in the North American Opiate Medication Initiative clinical trial. Addict Sci Clin Pract. 2014 Sep 29;9(1):21. doi: 10.1186/1940-0640-9-21. PMID 25262567
- [Derived] Oviedo-Joekes E, Guh D, Marchand K, Marsh DC, Lock K, Brissette S, Anis AH, Schechter MT. Differential long-term outcomes for voluntary and involuntary transition from injection to oral opioid maintenance treatment. Subst Abuse Treat Prev Policy. 2014 Jun 8;9:23. doi: 10.1186/1747-597X-9-23. PMID 24908387
- [Derived] Marchand K, Oviedo-Joekes E, Guh D, Marsh DC, Brissette S, Schechter MT. Sex work involvement among women with long-term opioid injection drug dependence who enter opioid agonist treatment. Harm Reduct J. 2012 Jan 25;9:8. doi: 10.1186/1477-7517-9-8. PMID 22276954
- [Derived] Marchand KI, Oviedo-Joekes E, Guh D, Brissette S, Marsh DC, Schechter MT. Client satisfaction among participants in a randomized trial comparing oral methadone and injectable diacetylmorphine for long-term opioid-dependency. BMC Health Serv Res. 2011 Jul 26;11:174. doi: 10.1186/1472-6963-11-174. PMID 21791093
- [Derived] Oviedo-Joekes E, Brissette S, Marsh DC, Lauzon P, Guh D, Anis A, Schechter MT. Diacetylmorphine versus methadone for the treatment of opioid addiction. N Engl J Med. 2009 Aug 20;361(8):777-86. doi: 10.1056/NEJMoa0810635. PMID 19692689
- [Derived] Gartry CC, Oviedo-Joekes E, Laliberte N, Schechter MT. NAOMI: The trials and tribulations of implementing a heroin assisted treatment study in North America. Harm Reduct J. 2009 Jan 21;6:2. doi: 10.1186/1477-7517-6-2. PMID 19159475
- See also: Related Info — http://www.naomistudy.ca